CLINICAL TRIAL: NCT00630357
Title: A Phase IV, Open-label, Multi-center Trial to Evaluate the Safety and Efficacy of Keppra® After Conversion to Mono-therapy in Adult Subjects With Partial Epilepsy
Brief Title: Trial to Evaluate the Safety and Efficacy of Keppra After Conversion to Mono-therapy in Subjects With Partial Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Study Director, UCB
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01037
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2009-09

CONDITIONS: Epilepsy
Keywords: Levetiracetam; Keppra
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levetiracetam (Keppra)

SUMMARY:
A cohort of patients who became seizure-free during add-on treatment to one standard AED with Keppra in a previous trial (N01031) were followed to assess whether seizure freedom was maintained. Tolerability was documented.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy with partial seizures;
* having completed the trial N01031 of Keppra as adjunctive therapy (SKATE);
* seizure-free over the last 3 months prior to protocol Visit 1;
* 1 concomitant marketed AED at the time of trial entry and throughout the previous trial N01031;
* on the clinical judgment of the Investigator, progressive withdrawal of the concomitant AED and conversion to monotherapy with Keppra can be attempted.

Exclusion Criteria:

* History of suicide attempt, current suicidal ideation, or other serious psychiatric disorders requiring or having required hospitalization or medication within the previous 5 years;
* presence of known pseudoseizures within the last year;
* presence or history of allergy to the components of Keppra (levetiracetam, lactose, cornstarch, and excipients) or other pyrrolidine derivatives;
* felbamate with less than 18 months exposure;
* vigabatrin, without visual field assessment as per recommendation of the manufacturer, i.e., every 6 months;
* uncountable seizures (clusters) or history of convulsive status epilepticus within the last 5 years.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2003-03; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Investigate seizure freedom with Keppra flexible dose.

SECONDARY OUTCOMES:
Tolerability and safety.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)